CLINICAL TRIAL: NCT02517216
Title: Parabolic Flight Induced Neuroplasticity Studied With Advanced Magnetic Resonance Imaging Methods
Acronym: BrainDTI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-004
Record Dates: First submitted 2015-07-21; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- parabolic flight and MRI scans (Other)
  Interventions: Other: parabolic flight; Device: MRI

INTERVENTIONS:
Other: parabolic flight
Device: MRI

SUMMARY:
Weightlessness profoundly modifies many physiological systems and especially the nervous system and the vestibular system. The changes in the nervous system are based in part on brain plasticity mechanisms, that is to say on modifications of neurons and their connections. They are the source of some of the behavioral response observed in the parabolic flight or in astronauts. For example, it is commonly observed that in the second and third days of parabolic flight campaigns with 3 flights, fewer participants are prone to motion sickness during the first day. Similarly, during their first trip into space, astronauts suffer 2/3 for 2 or 3 days of space sickness - special form of motion sickness - while this proportion is much lower in the second trip.

The hypothesis of this study is that short-term weightlessness as well as changes in the level of gravity experienced during parabolic flights, induce neuroplascity phenomena in brain regions involved in the integration of vestibular, visual and proprioceptive.

The goal is to objectify these plasticity phenomena, and assess their changes over time, using methods of Magnetic Resonance Imaging (MRI). A standard MRI will give an anatomical image of the brain. For this study, a variant called diffusion MRI (Diffusion Tensor Imaging - DTI) will visualize nerve bundles and their journey in the brain. The total duration of this review will be about ¾ hour.

The results of this study will be compared with those of an ongoing study of 12 astronauts who have the same MRI scans taken before and after a trip to the International Space Station. Investigators can then evaluate the effect of duration of exposure to weightlessness on the phenomena of neuroplasticity.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy volunteers (men or women)

  * Aged from 21 to 65
  * Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
  * Who accepted to take part in the study
  * Who have given their written stated consent
  * Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude. There will be no additional test performed for subject selection.
  * Who has already been included in the Belgium part of this experiment and thus has signed the Belgium informed consent.

Exclusion Criteria:

* • Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated

  * Person who has participated in a parabolic flight in the 2 previous years
  * Person with medical history of claustrophobia
  * Person with countraindication to MRI
  * Pregnant women

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
biomarkers of neuroplasticity with MRI | change over baseline and 6 months
  to identify biomarkers of neuroplasticity in the brain by comparing images before and after parabolic flight using advanced MRI methods
time course of possible changes and signs of neuroplasticity with MRI | change over baseline and 6 months
motion sickness questionnaires | change over baseline and 6 months
  to link biomarkers of brain plasticity with clinical outcome - obtained by motion sickness questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France